CLINICAL TRIAL: NCT04452929
Title: The Effect of Anti-calcitonin Gene-related Peptide (CGRP) Receptor Antibodies on the Headache Inducing Properties of CGRP and Cilostazol in Migraine Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Messoud Ashina, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CGRP2020
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Migraine; Migraine Without Aura; Migraine With Aura
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura | interventions — erenumab; Calcitonin Gene-Related Peptide; Cilostazol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, parallel study followed by a 6-month open-label extension.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized treatment phase: Erenumab (Active Comparator): Erenumab 140 mg single subcutaneous injection at baseline
  Interventions: Drug: Erenumab; Drug: Calcitonin gene-related peptide; Drug: Cilostazol
- Randomized treatment phase: Placebo (Placebo Comparator): Saline placebo single subcutaneous injection at baseline
  Interventions: Drug: Placebo; Drug: Calcitonin gene-related peptide; Drug: Cilostazol
- Open-label extension treatment phase: Erenumab (Other): Erenumab 140 mg monthly subcutaneous injection for six months after completion of the randomized, double-blinded, placebo-controlled study phase during the open-label extension
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Subcutaneous injection of 140 mg erenumab.
  Other Names: Aimovig®
  Arms: Open-label extension treatment phase: Erenumab; Randomized treatment phase: Erenumab
Drug: Placebo — Subcutaneous injection of saline placebo.
  Other Names: Saline placebo
  Arms: Randomized treatment phase: Placebo
Drug: Calcitonin gene-related peptide — Intravenous infusion of 1.5ug/min calcitonin gene-related peptide over 20 minutes.
  Arms: Randomized treatment phase: Erenumab; Randomized treatment phase: Placebo
Drug: Cilostazol — Oral intake of 200 mg cilostazol.
  Arms: Randomized treatment phase: Erenumab; Randomized treatment phase: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel study to investigate the effect of erenumab in calcitonin-gene related peptide and cilostazol experimental models of migraine in humans. Followed by a 6-month open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraine with or without aura according to the International Classification of Headache Disorders with a frequency of ≥4 migraine days per month
* 50-100 kg weight
* Participants of childbearing potential must use safe contraception (birth control) or be sexually abstinent

Exclusion Criteria:

* Any other primary headache disorder according to the International Classification of Headache Disorders except for tension-type headache
* Any secondary headache disorder according to the International Classification of Headache Disorders
* Migraine attack during the preceding 48 hours on provocation day
* Headache during the preceding 24 hours on provocation day
* Treatment with monoclonal antibodies or participation in clinical trials with monoclonal antibodies during the preceding year
* Daily consumption of any other drug/medication than oral contraception (birth control)
* Consumption of any other drug/medication later than four times the plasma half-time of the drug on provocation day except for oral contraception
* Pregnant or active breastfeeding participants
* Any cardiovascular diseases including cerebrovascular disorders
* Information in patient history or during physical examination indicating psychiatric disorders or substance abuse
* Information in patient history or during physical examination that the screening physician deems relevant for participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Migraine-like attack | Before (-5 min) and after administration of (+12 hours) of experimental trigger
  The incidence of migraine-like attack after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
  A migraine-like attack is defined attack fulfilling either (i) or (ii):
  (i) Headache fulfilling criteria C and D for migraine without aura according to the International Headache Society criteria: C. Headache has at least two of the following characteristics: unilateral location; pulsating quality; moderate or severe pain intensity (moderate to severe pain intensity is considered ≥4 on verbal rating scale); aggravation by cough (in-hospital phase) or causing avoidance of routine physical activity (out-hospital phase); D. During headache at least one of the following: nausea and/or vomiting; photophobia and phonophobia; and (ii) Headache described as mimicking the patient's usual migraine attack and treated with acute migraine medication (rescue medication).

SECONDARY OUTCOMES:
Headache intensity | Before (-5 min) and after administration of (+12 hours) of experimental trigger
  Change in headache intensity after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no pain; 10 is the worst pain imaginable.
Hemodynamics (superficial temporal artery) | Before (-5 min) and after administration of (+90 minutes) of experimental trigger
  Change in diameter (mm) of superficial temporal artery after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
Hemodynamics (radial artery) | Before (-5 min) and after administration of (+90 minutes) of experimental trigger
  Change in diameter (mm) of radial artery after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
Neuropeptide plasma concentrations (CGRP) | (1) Before (-5 min) and after administration of (+60 minutes) of experimental trigger; (2) 24-week open-label treatment phase
  1. Change in plasma concentrations of calcitonin gene-related peptide (CGRP) after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
  2. Change in plasma concentrations of calcitonin gene-related peptide during the open-label treatment phase.
Neuropeptide plasma concentrations (VIP) | (1) Before (-5 min) and after administration of (+60 minutes) of experimental trigger; (2) 24-week open-label treatment phase
  1. Change in plasma concentrations of vasoactive intestinal peptide (VIP) after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
  2. Change in plasma concentrations of vasoactive intestinal peptide (VIP) during the open-label treatment phase.
Neuropeptide plasma concentrations (PACAP) | (1) Before (-5 min) and after administration of (+60 minutes) of experimental trigger; (2) 24-week open-label treatment phase
  1. Change in plasma concentrations of pituitary adenylate cyclase-activating peptide (PACAP) after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
  2. Change in plasma concentrations of pituitary adenylate cyclase-activating peptide (PACAP) during the open-label treatment phase.
Facial flushing | Before (-5 min) and after administration of (+90 minutes) of experimental trigger
  Change in facial skin flushing after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
Facial temperature | Before (-5 min) and after administration of (+90 minutes) of experimental trigger
  Change in facial temperature after administration of calcitonin-gene related peptide or cilostazol in patients with migraine pretreated with erenumab compared to patients with migraine pretreated with placebo.
Headache day | Baseline and the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase
  Change in number of headache days per month after administration of erenumab from baseline compared to the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase.
Migraine day | Baseline and the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase
  Change in number of migraine days per month after administration of erenumab from baseline compared to the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase.
≥50% responder rate | Baseline and the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase
  Proportion of participants with a ≥50% reduction in number of migraine days per month after administration of erenumab from baseline compared to the last 3 months (months 4, 5, and 6) of the 24-week open-label treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Thien P Do, MD, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No